CLINICAL TRIAL: NCT06523101
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of PJ009 in Healthy Adult Volunteers
Brief Title: A Study of PJ009 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Peg-Bio Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQPJ-PJ009-001
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PJ009 group (Experimental): Participants will receive a single dose of PJ009 on day1, and then multiple doses of PJ009 once daily for 7 days (day5-11). Three dose levels will be evaluated. subcutaneous injection
  Interventions: Drug: PJ009
- PJ009 Placebo group (Placebo Comparator): Participants will receive a single dose of PJ009 placebo on day1, and then once daily for 7 days (day5-11). subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PJ009 — Six participants in each dose level will be randomized to receive a single dose and/or multiple doses of PJ009 in a double-blind fashion.
  Other Names: Glucagon-like Peptide-2 (GLP-2) analogue
  Arms: PJ009 group
Drug: Placebo — Two participants in each dose level will be randomized to receive placebo in a double-blind fashion.
  Arms: PJ009 Placebo group

SUMMARY:
The main aim of this clinical trial is to assess the safety of PJ009 in healthy adult volunteers aged 18-45. The main questions it aims to answer are:

* Is PJ009 safe in healthy adult? Participants will
* Receive single dose of PJ009 or placebo according to weight, and then multiple doses daily for 7 days,
* Stay in hospital for assessment.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, placebo-controlled phase 1 clinical study, aiming to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of PJ009 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign the informed consent form;
2. Healthy male or female subjects;
3. Aged 18 to 45 years (inclusive), body weight ≥ 50kg; body mass index between 19.0 and 26.0 (inclusive), body mass index (BMI) = weight (kg)/height^2 (m^2);
4. Female subjects of childbearing age with negative serum pregnancy test results;
5. Eligible subjects of fertility must agree to use effective contraceptive measures or abstain from sex during the study and within 6 months after the study;
6. Be able to understand and comply with the requirements of the protocol and expected to complete the entire study process.

Exclusion Criteria:

1. History of allergic diseases (including but not limited to asthma, urticaria, allergic rhinitis), drug allergy, or allergy to the ingredients of the investigational drug;
2. Used any drugs (including prescription drugs, over-the-counter drugs and Chinese herbal medicines) within 4 weeks before enrollment, except for external drugs that are not absorbed by the body; or used drugs known to cause significant damage to a certain organ within 12 weeks before enrollment;
3. History of any serious disease, including but not limited to digestive system, cardiovascular system, respiratory system, urinary system, musculoskeletal system, endocrine system, neuropsychiatric system, blood system, immune system diseases and metabolic abnormalities, or neurological or mental disorders, such as epilepsy and dementia;
4. History of congenital hemolytic hyperbilirubinemia;
5. History of gallstones or gastrointestinal surgery;
6. History of colorectal cancer;
7. History of gastrointestinal diseases, such as malabsorption, Crohn's disease, etc;
8. History of rash or dermatitis;
9. The laboratory and auxiliary examination results meet any of the following conditions:

   1. Abnormal electrocardiogram with clinical significance determined by the investigator;
   2. Abnormal vital signs with clinical significance determined by the investigator;
   3. Positive results of HIV-Ab, HCV-Ab, HBsAg or syphilis test;
   4. Abnormal results of laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function) with clinical significance;
   5. Positive results of drug abuse or alcohol test;
   6. Abnormal results of chest X-ray (anterior) with clinical significance determined by the investigator;
10. History of donating blood ≥ 200 mL within 12 weeks before enrollment, or plan to donate blood during the study;
11. History of major surgery within 12 weeks before enrollment;
12. History of alcohol abuse within 6 months before enrollment, that is, drinking more than 14 units of alcohol per week (1 unit = 12 ounces or 360 mL of beer, 1.5 ounces or 45 mL of liquor with an alcohol content of 40%, 5 ounces or 150 mL wine);
13. Smoke more than 5 cigarettes a day within 6 months before enrollment;
14. Participated in other clinical trials within 12 weeks before enrollment, or used similar drugs of the investigational drug;
15. Cannot tolerate venipuncture blood collection or have a history of needle or blood fainting;
16. Lactating, pregnant, or planning to become pregnant or conceive in the near future;
17. Poor compliance as assessed by the investigator;
18. The investigator believes the subject is unsuitable for participating in this clinical study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Treatment-related Adverse Events | Up to 18 days
  Number of participants with treatment-related adverse events during the study will be collected and the percentage of adverse events (AEs) of different grades as assessed by CTCAE v5.0 will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ruigang Hou, Principal Investigator — Second Hospital of Shanxi Medical University
Locations (1):
- The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi, China